CLINICAL TRIAL: NCT05845879
Title: Obstetrical Outcomes for Planned Deliveries in a French Birth Center
Acronym: NidaModa
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Matthieu DAP, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2022PI173
Record Dates: First submitted 2023-04-09; First posted 2023-05-06 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Delivery Complication
MeSH Terms: interventions — Parturition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women who planned to deliver at the brith center "un nid pour naître": Women who planned to deliver at the brith center "un nid pour naître"
  Interventions: Other: delivery

INTERVENTIONS:
Other: delivery — delivery

SUMMARY:
The main objective of this work is to study the obstetrical and neonatal outcomes of women who planned to deliver in the birth centre of Nancy.

The birth centre of Nancy is one of the nine french birth centres opened since 2015 on an experimental basis.

The women who plan to deliver at the birth centre must meet several conditions according to their medical history, pregnancy follow-up, and delivery progress.

The women can be transferred before, during or after (pre-, per- or post-) delivery to the hospital.

ELIGIBILITY:
Inclusion Criteria:

* women who want to deliver at the birth center "Un nid pour naître"

Exclusion Criteria:

* Refusal to participate in the study.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: All women who want to deliver at the birth center "Un nid pour naître" since 01/01/2020 to 31/12/2022
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the cesarean birth rate of women who planned to deliver in the birth centre according to the final place of labor (hospital or birth centre). | 4 years
  rate of cesarean section
Comparison of the instrumental birth rate of women who planned to deliver in the birth centre according to the final place of labor (hospital or birth centre). | 4 years
  rate of instrumental birth (vacuum or forceps delivery)
Comparison of the post-partum haemorrhage rate of women who planned to deliver in the birth centre according to the final place of labor (hospital or birth centre). | 4 years
  rate of post-partum haemorrhage define by blood loss >= 500 cc

SECONDARY OUTCOMES:
Comparison of the antepartum or peripartum stillbirth rate of women who planned to deliver in the birth center according to the final place of labor (hospital or birth centre). | 4 years
Comparison of the hypoxemic encephalopathy rate of women who planned to deliver in the birth center according to the final place of labor (hospital or birth centre). | 4 years
Comparison of the five-minute Apgar score of babies from women who planned to deliver in the birth centre according to the final place of labor (hospital or birth centre). | 4 years
  Apgar score is a score that records the physical condition of a baby just after it is born, with ten points being the highest possible score and zero point the lowest.
Comparison of the umbilical artery blood pH score of babies from women who planned to deliver in the birth centre according to the final place of labor (hospital or birth centre). | 4 years